CLINICAL TRIAL: NCT04304287
Title: The Benefit of Autologous Blood Transfusion in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Zrinka Oreskovic, Principal investigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Orthopedia/autotransfusion
Record Dates: First submitted 2020-02-27; First posted 2020-03-11 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Transfusion; Hip Arthroplasty
Keywords: total hip arthroplasty; autologous blood donation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Preoperative blood donations 14 day before total hip replacement procedure Donation of one dose of autologous blood 14 day before total hip replacement procedure
  Interventions: Procedure: Preoperative autologous blood donation, 14 days before surgery
- Active comparator (Active Comparator): Preoperative blood donation 72 hours before total hip replacement procedure Donation of one dose of autologous blood 72 hours before total hip replacement procedure
  Interventions: Procedure: Preoperative autologous blood donation, 72 hours before surgery
- Other (Other): Without preoperative blood donation
  Interventions: Procedure: Without preoperative blood donation

INTERVENTIONS:
Procedure: Preoperative autologous blood donation, 14 days before surgery
  Arms: Experimental
Procedure: Preoperative autologous blood donation, 72 hours before surgery
  Arms: Active comparator
Procedure: Without preoperative blood donation
  Arms: Other

SUMMARY:
The investigators studied the benefit of preoperative autologous blood donation in participants who undergo total hip arthroplasty. Study is made as a prospective and randomized.

DETAILED DESCRIPTION:
Total hip arthroplasty is procedure followed with large perioperative and postoperative blood loss. In order to avoid the application of large amounts of allogeneic blood, preoperative autologous blood donation as a tipe of autologous transfusion have been developed.

In this study, the investigators studied the benefit of preoperative autologous blood donation in participants who undergo total hip arthroplasty. Study is made as a prospective and randomized.

Participants were divided into three groups: the first group donated one dose of autologous blood 14 days preoperatively, the second group donated one dose of autologous blood 72 hours preoperatively and a third group was not donated autologous blood.

The blood parameters, hemodynamic stability, bleeding, the need for application of autologous or homologous blood and length of hospital stay were compared.

ELIGIBILITY:
Inclusion Criteria:

* subject older than 18 years
* subject has primary coxarthrosis
* subject has indication for total hip replacement

Exclusion Criteria:

* subject has secondary coxarthrosis
* subject has need for revision endoprosthesis
* history of autoimmune, malignancy or coagulation disorder
* history of myocardial infarct or cerebrovascular insult in last 6 months
* history of angina pectoris and unregulated hypertension
* history of renal or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-01-16 (Actual); Primary Completion 2013-06-15 (Actual); Study Completion 2015-06-15 (Actual)

PRIMARY OUTCOMES:
Patient red blood cells value | 6 days
  analysis of blood sample day before surgery, 3 hours after surgery, on first, second, fifth postoperative day and on sixth postoperative day
Need for autologous blood transfusion | 6 days
  Based on blood count and hemodynamic stability
Need for homologous blood transfusion | 6 days
  Based on blood count and hemodynamic stability
Patient hemoglobin value | 6 days
  analysis of blood sample day before surgery, 3 hours after surgery, on first, second, fifth postoperative day and on sixth postoperative day
Patient hematocrit value | 6 days
  analysis of blood sample day before surgery, 3 hours after surgery, on first, second, fifth postoperative day and on sixth postoperative day

SECONDARY OUTCOMES:
Length of hospital stay | 6 days
  measure of length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Domagoj Delimar, MD, Study Director — Clinical Hospital Centre Zagreb

IPD SHARING:
Plan to Share IPD: No